CLINICAL TRIAL: NCT04395664
Title: The ACOVID-19 Study - A Prospective Cohort Study Investigating the Acute Effect of COVID-19 on the Heart by Continuous ECG Monitoring
Brief Title: Arrhythmias in Patients With COVID-19
Acronym: ACOVID
Status: Completed | Type: Observational
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Morten Lamberts, Associate Professor and Research Director, Herlev and Gentofte Hospital
Other Study IDs: H-20021500
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: C3+ Holter Monitor — ECG monitoring

SUMMARY:
The study is a prospective clinical cohort study of consecutive patients hospitalized at all hospitals of greater Copenhagen with a laboratory confirmed diagnosis of COVID-19. The investigators aim to examine if continuous ECG monitoring can be used to understand the contribution of COVID-19 infection in the acute phase to the development of cardiac arrhythmias, especially focusing on cardiovascular outcomes. In all patients included, the investigators aim to examine if continuous ECG monitoring - alone and in combination with biomarkers - can be used to detect early signs of cardiac complications and predict long-term risk of cardiovascular morbidity and mortality following COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized at hospitals of greater Copenhagen area and Zealand with a laboratory confirmed diagnosis of COVID-19 > 18 years of age.

Exclusion Criteria:

* Persons not able to cooperate
* Persons unable to understand and sign "informed consent"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In.patients from hospitals of the greater Copenhagen area
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality during hospitalization and a confirmed COVID-19 diagnosis | 4 months
Incident intensive care unit admission during hospitalization and a confirmed COVID-19 diagnosis | 4 months

SECONDARY OUTCOMES:
Incident pulmonary embolism during hospitalization and a confirmed COVID-19 diagnosis | 4 months
Incident cardiac arrest during hospitalization and a confirmed COVID-19 diagnosis | 4 months
Incident hypoxic respiratory failure during hospitalization and a confirmed COVID-19 diagnosis | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Herlev & Gentofte Hospital, Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided